CLINICAL TRIAL: NCT00606944
Title: Randomized Controlled Trial of Fast-Track Rehabilitation After Elective Colorectal and Small Bowel Resection
Brief Title: Fast-track Rehabilitation After Elective Colorectal and Small Bowel Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sung-Bum Kang, Associate Professor Department of Surgery, Seoul National University Bundang Hospita, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-0706-046-008; SNUBH-GS-CR1
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-07

CONDITIONS: Colorectal Tumor
Keywords: enhanced recovery program
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ERP group (Experimental): fast-track rehabilitation with early ambulation and diet after elective colorectal resection
  Interventions: Behavioral: fast-track rehabilitation
- control group (No Intervention): traditional, conventional care group

INTERVENTIONS:
Behavioral: fast-track rehabilitation — fast-track rehabilitation with early ambulation and diet after elective colorectal resection
  Arms: ERP group

SUMMARY:
The purpose of this study is to address the question of whether or not oral alimentation and ambulation exercise should be begun early in patients following laparoscopic colorectal surgery compared to the classical diet and ambulation which depends on reappearance of functional intestinal transit. Early oral alimentation following laparoscopic colorectal surgery may decrease hospital stay and facilitate earlier discharge with comparable postoperative morbidity.

DETAILED DESCRIPTION:
Traditionally, patients who received laparoscopic colorectal surgery were treated with the classical protocol including the use of a naso-gastric tube and starvation for several postoperative days till the recovery of bowel movement, or bed resting at immediate postoperative period followed by ward ambulation at the postoperative day 1 or 2. Restarting the oral alimentation is based on gas or feces reappearance after surgery and usually this is possible at several days following surgery. However, prolonged starvation might be uncomfortable for the patient as well as increasing his postoperative hospital stay. Recently, several studies reported the efficacy of early rehabilitation protocols after intestinal surgery, showing that early oral alimentation could reduce the length of hospital stay and cost of hospitalization without significant increase of postoperative complications, compared to traditional management.

This prospective, randomized study was designed to evaluate the effectiveness of a postoperative care pathway using rehabilitation with early ambulation and diet for patients undergoing elective laparoscopic colorectal resection compared with the traditional postoperative care.

In order to conduct this study, patients having a laparoscopic colon resection will be randomly attributed to enhanced recovery program group or control group, which is divided based on the postoperative management protocol.

ELIGIBILITY:
Inclusion Criteria:

* • Patients between 20 - 80 years old

  * Class ASA (American Society of Anesthesiology) I, II or III, +/- E
  * Patient willing to participate in the study
  * Patient who understands and accepts to sign the informed consent form
  * Patient who will undergo elective colorectal resection using laparoscopic surgery defined as follows: patients who received one of the following surgery:right hemicolectomy, left hemicolectomy, anterior resection with primary anastomosis, and low anterior resection with loop ileostomy for fecal diversion

Exclusion Criteria:

* • Class ASA IV or V patient

  * Documented problem of gastro-intestinal motility
  * Combined resection of other organ than the colorectum
  * Presence of obstructive colorectal cancer associated with dilatation of the proximal gastrointestinal tract
  * Presence of residual peritoneal carcinosis at the end of surgery
  * Previous history of intra-abdominal surgery except simple appendectomy, cholecystectomy, or hysterectomy for uterine myoma
  * Creation of colo-rectal, colo-anal or ileo-anal anastomosis without loop ileostomy
  * Any per-surgery discovery which requires the use of a gastric drainage procedure following surgery
  * Any post-surgery change in patient condition which requires naso-gastric tube holding after surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-06; Primary Completion 2009-10 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bum Kang, M.D., Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Department of Surgery, Seoul National University Bundang Hospital, Seongnam
  - Sung-Bum Kang, Seongnam

REFERENCES:
- [Derived] Lee SM, Kang SB, Jang JH, Park JS, Hong S, Lee TG, Ahn S. Early rehabilitation versus conventional care after laparoscopic rectal surgery: a prospective, randomized, controlled trial. Surg Endosc. 2013 Oct;27(10):3902-9. doi: 10.1007/s00464-013-3006-4. Epub 2013 May 25. PMID 23708720
- [Derived] Lee TG, Kang SB, Kim DW, Hong S, Heo SC, Park KJ. Comparison of early mobilization and diet rehabilitation program with conventional care after laparoscopic colon surgery: a prospective randomized controlled trial. Dis Colon Rectum. 2011 Jan;54(1):21-8. doi: 10.1007/DCR.0b013e3181fcdb3e. PMID 21160309

RESULTS

PARTICIPANT FLOW:
Groups:
- ERP Group: Early rehabilitation program after laparoscopic colorectal surgery with early oral alimentation and early ambulation
Period: Overall Study
Arm/Group | Control Group | ERP Group
Started | 98 | 100
Completed | 98 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ERP Group: Early rehabilitation program after laparoscopic colon surgery with early oral alimentation and early ambulation
- Total: Total of all reporting groups
Arm/Group | Control Group | ERP Group | Total
Number analyzed (Participants) | 100 | 98 | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 49 | 107
  >=65 years | 42 | 49 | 91
Age Continuous [Mean (Standard Deviation); unit: years] | 61.1 (11.0) | 61.5 (10.9) | 61.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 36 | 78
  Male | 58 | 62 | 120
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 100 | 98 | 198

OUTCOME MEASURES:

1. Primary Outcome: the Length of Hospital Stay
Description: discharge criteria
  1. Tolerance of consecutive 3 soft bland diet
  2. Unassisted ambulation
  3. No necessity of analgesics
  4. Afebrile without major complication
  5. Willing to discharge
Time Frame: at discharge
Population: 1 mortality case was excluded for analysis in the ERP group
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Control Group | ERP Group
Number analyzed (Participants) | 100 | 97
day | 8 [7 to 9] | 7 [6.75 to 8.25]

2. Primary Outcome: Pain
Description: score measured by the Visual Analog Scale
Time Frame: at discharge
Reporting Status: Not Posted

3. Primary Outcome: Quality of Life
Description: measured by SF-36
Time Frame: at discharge
Reporting Status: Not Posted

4. Primary Outcome: Postoperative Complication During the First Admission
Time Frame: at discharge
Reporting Status: Not Posted

5. Primary Outcome: Recovery
Description: recovery criteria must include all of the following
  1. Tolerance of consecutive 3 soft bland diet
  2. Unassisted ambulation
  3. No necessity of analgesics
  4. Afebrile without major complication
Time Frame: at discharge
Reporting Status: Not Posted

6. Secondary Outcome: Readmission Rate
Time Frame: at postoperative day 30
Reporting Status: Not Posted

7. Secondary Outcome: Pain
Description: score measured by the Visual Analog Scale
Time Frame: at postoperative day 30
Reporting Status: Not Posted

8. Secondary Outcome: Quality of Life
Description: measured by SF-36
Time Frame: at postoperative day 30
Reporting Status: Not Posted

9. Secondary Outcome: Postoperative Complication
Time Frame: at postoperative day 30
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Control Group | ERP Group
Serious Adverse Events (participants affected / at risk) | 0/100 | 1/98
Other Adverse Events (participants affected / at risk) | 16/100 | 28/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=100) | ERP Group (N=98)
Death (Gastrointestinal disorders) | 0 (0) | 1 (1) — 1 patient in ERP group who underwent low anterior resection for rectal cancer died due to aspiration pneumonia at postoperative 3day
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=100) | ERP Group (N=98)
Ileus (Gastrointestinal disorders) | 7 (7) | 17 (17) — defined by patient's symptom and X-ray
Urinary retention (Renal and urinary disorders) | 5 (5) | 9 (9)
Chylous ascites (Gastrointestinal disorders) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No